CLINICAL TRIAL: NCT01736462
Title: An Open-Label Study to Evaluate 3 Month Corneal Endothelial Cell Density Changes in Healthy Subjects When Mapracorat Ophthalmic Suspension, 3%, is Administered 4 Times Daily for 14 Days
Brief Title: Corneal Endothelial Cell Density Changes, When Mapracorat Ophthalmic Suspension 3%, is Administered for 14 Days
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 794
Record Dates: First submitted 2012-11-20; First posted 2012-11-29 (Estimated); Last update posted 2013-11-26 (Estimated); Status verified 2013-11

CONDITIONS: Corneal Endothelial Cell Changes
Keywords: Cornea; Endothelial cell density
MeSH Terms: conditions — Corneal Diseases | interventions — R-1,1,1-trifluoro-4-(5-fluoro-2,3-dihydrobenzofuran-7-yl)-4-methyl-2-(((2-methyl-5-quinolyl)amino)methyl)pentan-2-ol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mapracorat (Experimental): Mapracorat ophthalmic suspension, 3%
  Interventions: Drug: Mapracorat

INTERVENTIONS:
Drug: Mapracorat — One drop of mapracorat ophthalmic suspension, 3% four times daily, at approximately four hour intervals, for 14 days in both eyes.

SUMMARY:
The objective of this study is to evaluate the effect on corneal endothelial cell density (cells/mm²) changes at 3 months when mapracorat ophthalmic suspension, 3% is administered QID (four times daily), for 14 days in healthy subjects with a normal ophthalmic history.

ELIGIBILITY:
Inclusion Criteria:

* Must have a Pinhole visual acuity (VA) equal to or better than 20/40 in both eyes.
* Must be in good ocular health

Exclusion Criteria:

* Subjects who have known hypersensitivity or contraindication to the study drug or its components.
* Subjects who currently require or are expected to require treatment with any medication listed as a disallowed medication per the Disallowed Therapy section of the protocol.
* Any topical ophthalmic medication, including tear substitutes that cannot be discontinued during the study.
* Subjects who are monocular (fellow eye is absent or fellow eye's Pinhole VA is worse than 20/200).
* Subjects with a history of ocular surgery, or who anticipate ocular surgery in either eye within the study period.
* Presence of significant ocular or systemic disease that the Investigator determines could interfere with the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2013-02; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Endothelial Cell Density | 3 months (Visit 4)
  The mean endothelial cell density (cells/mm2)(ECD)

SECONDARY OUTCOMES:
Area under the plasma concentration-time curve | Day 1 (Visit 2)
  Area under the plasma concentration-time curve from time 0 to the time of the last quantifiable concentration (Ct). Blood samples will be collected for the determination of mapracorat and any potential metabolite(s). Concentrations in plasma measured within 1 hour prior to dosing on day 1 (visit 2).
Area under the plasma concentration-time curve | Day 15 (Visit 3)
  Area under the plasma concentration-time curve from time 0 to the time of the last quantifiable concentration (Ct). Blood samples will be collected for the determination of mapracorat and any potential metabolite(s). Blood samples will be collected within 1 hour prior to dosing and at 0.25, 0.5, 1, 2, and 4 hours after a single administration of mapracorat at visit 3.

CONTACTS AND LOCATIONS:
Overall Officials: Quintus Ngumah, OD, PhD, Study Director — Bausch & Lomb Incorporated
Locations (1):
- Bausch & Lomb Inc, Rochester, New York, United States